CLINICAL TRIAL: NCT03955289
Title: Treatment of Foot and Leg Ulcers Using a Laser
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Larry Lavery, Professor and Director of Research, University of Texas Southwestern Medical Center
Other Study IDs: 2018-0270
Record Dates: First submitted 2019-05-16; First posted 2019-05-20 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators plan to do a retrospective chart review on patients who underwent laser treatment for their foot ulcer at the UT Southwestern wound clinic.

DETAILED DESCRIPTION:
The investigators plan to do a retrospective chart review on patients who underwent laser treatment for their foot ulcer at the UT Southwestern wound clinic starting on May 17, 2018 to November 13, 2018. The investigators chose this date because that is the first time laser treatments were performed in the clinic. The investigators will collect the following data points:

* Ulcer etiology
* Ulcer location
* Prior ulcer treatment type and duration, and wound measurements/characteristics
* Wound size 4-6 weeks prior to laser treatment; at treatment time; and then each follow up measurement healed or x weeks
* eGFR
* Albumin
* Last A1c-Presence/absence of DM
* Amputation history
* Vascular status via ABI's
* Identify comorbidities
* Identify associated encounters in the patients such as complications (i.e. infection), related readmissions The investigators will identify this information from patient charts (EPIC EMR).

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent laser treatment for their foot ulcer at the UT Southwestern wound clinic starting on May 17, 2018 to November 13, 2018

Exclusion Criteria:

* not meeting inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of the investigators with foot ulcers.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Improved healing rate to time to healing | 4 weeks
  Wounds assessed in this study will show significant improvement in wound characteristics after Erbium-YAG laser debridement(s). Improved healing rate to time to healing.

SECONDARY OUTCOMES:
Decreased complications in diabetic foot ulcers, i.e. infection, hospital admission, amputation | 4 weeks
  Wounds assessed in this study will show significant improvement in wound characteristics after Erbium-YAG laser debridement(s).
  Decreased complications in diabetic foot ulcers, i.e. infection, hospital admission, amputation

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Lavery, DPM MPH, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center at Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rice JB, Desai U, Cummings AK, Birnbaum HG, Skornicki M, Parsons NB. Burden of diabetic foot ulcers for medicare and private insurers. Diabetes Care. 2014;37(3):651-8. doi: 10.2337/dc13-2176. Epub 2013 Nov 1. PMID 24186882
- [Background] Teikemeier G, Goldberg DJ. Skin resurfacing with the erbium:YAG laser. Dermatol Surg. 1997 Aug;23(8):685-7. doi: 10.1111/j.1524-4725.1997.tb00389.x. PMID 9256915
- [Background] Mezzana P, Sonnino M, Madonna Terracina FS, Valeriani M. Treatment of atrophic scars with Er:YAG laser: our experience. Acta Chir Plast. 2001;43(1):26-8. PMID 11370255
- [Background] Wollina U, Konrad H, Karamfilov T. Treatment of common warts and actinic keratoses by Er:YAG laser. J Cutan Laser Ther. 2001 Jun;3(2):63-6. doi: 10.1080/146288301753377852. PMID 11798495
- [Background] Gurel MS, Aral BB. Effectiveness of erbium:YAG laser and cryosurgery in seborrheic keratoses: Randomized, prospective intraindividual comparison study. J Dermatolog Treat. 2015 Oct;26(5):477-80. doi: 10.3109/09546634.2015.1024597. Epub 2015 Mar 23. PMID 25798694
- [Background] Alsaad SM, Ross EV, Smith WJ, DeRienzo DP. Analysis of Depth of Ablation,Thermal Damage, Wound Healing, and Wound Contraction With Erbium YAG Laser in a Yorkshire Pig Model. J Drugs Dermatol. 2015 Nov;14(11):1245-52. PMID 26580873
- [Background] Madni TD, Lu KB, Imran JB, Clark AT, Hoopman JE, Kenkel JM, Phelan HA. Chronic burn wound treatment by Erbium: YAG fractional ablation: First described report and literature review. Burns. 2019 Feb;45(1):256-258. doi: 10.1016/j.burns.2018.10.001. Epub 2018 Oct 17. No abstract available. PMID 30342793
- [Background] Phillips TJ, Morton LM, Uebelhoer NS, Dover JS. Ablative Fractional Carbon Dioxide Laser in the Treatment of Chronic, Posttraumatic, Lower-Extremity Ulcers in Elderly Patients. JAMA Dermatol. 2015 Aug;151(8):868-71. doi: 10.1001/jamadermatol.2015.0645. PMID 25946007
- [Background] Krakowski AC, Diaz L, Admani S, Uebelhoer NS, Shumaker PR. Healing of chronic wounds with adjunctive ablative fractional laser resurfacing in two pediatric patients. Lasers Surg Med. 2016 Feb;48(2):166-9. doi: 10.1002/lsm.22398. Epub 2015 Aug 7. PMID 26251161
- See also: 2. Sciton Inc. (n.d.). [Brochure]. Author. Retrieved November 8, 2018 — https://sciton.com/physicians/profractional
- See also: Wollina, Uwe. (2016). Erbium-YAG laser therapy - analysis of more than 1,200 treatments. Journal of Global Dermatology. 3. 10.15761/GOD.1000171 — https://www.researchgate.net/publication/299493475_Erbium-YAG_laser_therapy_-_analysis_of_more_than_1200_treatments